CLINICAL TRIAL: NCT00670631
Title: Tandem Autotransplantation for Multiple Myeloma Patients With Less Than 12 Months of Preceding Therapy, Incorporating Bortezomib With the Transplant Chemotherapy and During Maintenance
Brief Title: Tandem Transplantation in Multiple Myeloma (MM) Patients With <12 Months of Prior Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guido Tricot (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Guido Tricot, Guido J.K. Tricot, MD, PhD, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25009; 7R01CA115399 (NIH)
Record Dates: First submitted 2008-04-03; First posted 2008-05-02 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Intervention Model Description: Induction- Tandem Transplants with VTD-MEL and gemcitabine, BCNU, melphalan, velcade and dexamethasone- Maintenance therapy
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tandem autologous stem cell transplant (Experimental): Induction: DPACE(dexamethasone,cisplatin,doxorubicin,cyclophosphamide,etoposide) chemotherapy plus stem cell collection. Additional stem cell collection and/or chemotherapy may be required.
  After collection, participants will receive dexamethasone x 4 days every 14 days.
  Transplant 1: The transplant preparative regimen will be bortezomib/thalidomide/dexamethasone/melphalan.
  Once recovered, participants start thalidomide daily and dexamethasone x 4 days every 21 days.
  Consolidation (if administered): VDT-PACE(bortezomib,dexamethasone,thalidomide,cisplatin,doxorubicin,cyclophosphamide, etoposide) Transplant 2: 8 weeks to 6 months after the first transplant, participants will have the second transplant Maintenance: Year 1- VTD (bortezomib, thalidomide, dexamethasone) cycles. Year 2 - VCD (bortezomib, cyclophosphamide, dexamethasone)cycles.
  Interventions: Combination Product: tandem autologous transplantation

INTERVENTIONS:
Combination Product: tandem autologous transplantation — DPACE: dexamethasone 20 mg days 1-4 and 8-11, cisplatin 10 mg/m2 days 1-4, Adriamycin 10 mg/m2 days 1-4, cyclophosphamide 400 mg/m2 days 1-4, etoposide 40 mg/m2 days 1-4.
  Transplant 1: Dexamethasone 20 mg days -4 to -1 and +2 to +5. Velcade 1mg/m2 on days -4,-1, +2, and +5. Thalidomide 100mg on day -4 to day +5. Melphalan, 100 mg/m2 on days -4 and -1.
  Transplant 2: Dexamethasone 20 mg on days -4 to -1 and +2 to +5. BCNU 300mg/m2 on day -4. Melphalan 140 mg/m2 on day -1. Velcade 1mg/m2 on days -4, -1, +2, +5. Gemcitabine 1000 mg/m2 on days -4 + -1.
  Maintenance year 1: Bortezomib 1.0 mg/m2 on days 1, 4, 15,18 every cycle. Thalidomide, 100 mg . Dexamethasone,20 mg,on days 1-4 & 15-18 every cycle.
  Maintenance year 2: Dexamethasone, 20 mg,days 1-4 every cycle.

SUMMARY:
The two objectives of this study are:

* To increase the 2-year event-free survival from 55%, established with Total Therapy II (UARK 98-026), to 75% in myeloma patients with cytogenetic abnormalities, and from 80%, established with the Total Therapy II regimen, to 95% in myeloma patients without cytogenetic abnormalities.
* To determine whether bortezomib, thalidomide, and dexamethasone can be safely incorporated with transplant 1 into the established pre-transplant regimen of high-dose melphalan (used in Total Therapy II) and whether Velcade and gemcitabine can be safely added to the transplant 2 high-dose chemotherapy regimen of combination melphalan and BCNU.

DETAILED DESCRIPTION:
This study is targeted towards patients who have been diagnosed with Multiple Myeloma and have had no prior autologous or allogeneic transplant. Furthermore, only up to 12 months of prior treatment are allowed in this patient population. The study schema consists of one round of induction chemotherapy, two transplants, one round of consolidation chemotherapy, and two years of maintenance treatment. This study design differs from its historical predecessors in the following manner:

* In contrast to Total Therapy II and III, which only allow enrollment of patients with at most one cycle or one month of treatment prior to enrollment, the proposed study allows enrollment of patients with up to 12 months of prior treatment. No statistically significant difference in outcome between patients with one or no cycle of preceding therapy and those with up to 12 months of prior therapy. This should allow enrollment of significantly more myeloma patients.
* Induction therapy has been reduced to a single cycle.
* Bortezomib and thalidomide have been added to the transplant regimen.
* BCNU is added to the second transplant to high dose melphalan.
* Gemcitabine is added to the second transplant regimen.
* Consolidation treatment has been reduced to a single cycle.
* The first year of maintenance is with bortezomib, thalidomide and dexamethasone, and the second year of maintenance therapy consists of dexamethasone only.
* The novel agents thalidomide and bortezomib are not introduced upfront, but only with transplantation and maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the diagnosis of active MM requiring treatment. Patients with a previous history of smoldering myeloma will be eligible if there is evidence of progressive disease requiring chemotherapy.
2. Protein criteria must be present (quantifiable M-component of IgG, IgA, IgD, or IgE and/or urinary kappa or lambda light chain, Bence-Jones protein, or Free Kappa Light Chain or Free Lambda Light Chain) in order to evaluate response. Non-secretory patients are eligible provided the patient has > 20% plasmacytosis OR multiple (>3) focal plasmacytomas or focal lesions on MRI.
3. Patients must have received no more than 12 months of prior chemotherapy for this disease. Patients may have received prior radiotherapy provided approval has been obtained by the Principal Investigator.
4. Patients must be 18-75 years of age at the time of initial registration.
5. Ejection fraction by ECHO or MUGA ≥ 40% performed within 60 days prior to registration.
6. Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, FVC) and diffusion capacity (DLCO) > 50% of predicted, within 60 days of registration. If the patient is unable to complete pulmonary function tests due to MM related pain or condition, exception may be granted if the principal investigator documents that the patient is a candidate for high dose therapy.
7. Patients must have a creatinine < 3 mg/dl and a creatinine clearance >30mL/min
8. Patients must have a performance status of 0-2 based on SWOG criteria. Patients with a poor performance status (3-4), based solely on bone pain will be eligible.
9. All patients must be informed of the investigational nature of this study and must have signed an IRB-approved informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

1. Platelet count < 30 x 109/L, unless myeloma-related.
2. Greater than a grade 2 peripheral neuropathy.
3. Hypersensitivity to bortezomib, boron, or mannitol.
4. Uncontrolled diabetes.
5. Recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias.
6. Evidence of chronic obstructive or chronic restrictive pulmonary disease.
7. Patients must not have light chain deposition disease-related renal failure or creatinine > 3 mg/dl.
8. Patients must not have prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will only be acceptable if the patient's life expectancy exceeds five years.
9. Patients must not have significant co-morbid medical conditions or uncontrolled life threatening infection.
10. Pregnant or nursing women. Women of child-bearing potential must have a negative pregnancy test documented within one week of registration. Women and men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-02; Primary Completion 2012-05 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido J Tricot, MD, PhD, Principal Investigator — University of Iowa

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data not available. Study conducted at University of Utah. Upon PI leaving Utah and coming to the University of Iowa, record NCT00670631 was transferred to Iowa by ClinicalTrials.gov staff. No research activities under NCT00670631 were conducted at Iowa. PRS staff at Iowa and Utah have corresponded and neither party (including PI) have the data.
Groups:
- Tandem Autologous Stem Cell Transplant: Induction: DPACE chemotherapy plus stem cell collection. Additional stem cell collection and/or chemotherapy may be required.
  After collection, participants will receive dexamethasone x 4 days every 14 days.
Period: Overall Study
Arm/Group | Tandem Autologous Stem Cell Transplant
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Data not available. Study conducted at University of Utah. Upon PI leaving Utah and coming to the University of Iowa, record NCT00670631 was transferred to Iowa by ClinicalTrials.gov staff. No research activities under NCT00670631 were conducted at Iowa. PRS staff at Iowa and Utah have corresponded and neither party (including PI) have the data.
Groups:
- Tandem Autologous Stem Cell Transplant: Induction: DPACE(dexamethasone,cisplatin,doxorubicin,cyclophosphamide,etoposide) chemotherapy plus stem cell collection. Additional stem cell collection and/or chemotherapy may be required.
  After collection, participants will receive dexamethasone x 4 days every 14 days.
Arm/Group | Tandem Autologous Stem Cell Transplant
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: To Determine Whether, in Comparison to TT II, the Median EFS Can be Increased From 4.8 Years to 6.2 Years, Which Represents an Increase in Median EFS of Approximately 30%
Time Frame: After enrollment of 204 subjects is completed
Population: as for baseline characteristics
Groups:
- Tandem Autologous Stem Cell Transplant: Induction: DPACE(dexamethasone,cisplatin,doxorubicin,cyclophosphamide,etoposide) chemotherapy plus stem cell collection. Additional stem cell collection and/or chemotherapy may be required.
  After collection, participants will receive dexamethasone x 4 days every 14 days.
  Transplant 1: The transplant preparative regimen will be bortezomib/thalidomide/dexamethasone/melphalan.
  Once recovered, participants start thalidomide daily & dexamethasone x 4 days every 21 days.
  Consolidation (if administered): VDT-PACE(bortezomib,dexamethasone,thalidomide,cisplatin,doxorubicin,cyclophosphamide, etoposide) Transplant 2: 8 weeks to 6 months after the first transplant, participants will have the second transplant Maintenance: Year 1- VTD (bortezomib, thalidomide, dexamethasone) cycles. Year 2 - VCD (bortezomib, cyclophosphamide, dexamethasone)cycles.
  tandem autologous transplantation: DPACE: dexamethasone 20 mg days 1-4 and 8-11, cisplatin 10 mg/m2 days 1-4, Adriamycin 10 mg/m2 days
Arm/Group | Tandem Autologous Stem Cell Transplant
Number analyzed (Participants) | 0

2. Primary Outcome: In Assessing Patient Safety, we Will Examine Treatment Toxicity Related Mortality and SAEs. Historical Study Results Indicate That a Mortality Rate of Greater Than 10% is Not Acceptable in This Population, Nor is an SAE Rate of Greater Than 15%.
Time Frame: Interim analyses for safety will be performed after 20, 100, 200, and 300 patients have been enrolled.
Population: as for baseline characteristics
Arm/Group | Tandem Autologous Stem Cell Transplant
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival Will be Compared to a Historical Control (UARK 98-026, TT2)as a Secondary Outcome.
Time Frame: After 204 patients have been enrolled
Population: as for baseline characteristics
Arm/Group | Tandem Autologous Stem Cell Transplant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Data not available. Study conducted at University of Utah. Upon PI leaving Utah and coming to the University of Iowa, record NCT00670631 was transferred to Iowa by ClinicalTrials.gov staff. No research activities under NCT00670631 were conducted at Iowa. PRS staff at Iowa and Utah have corresponded and neither party (including PI) have the data.
Arm/Group | Tandem Autologous Stem Cell Transplant
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Data not available. Study conducted at Utah. Upon PI leaving & coming to Iowa, record was transferred to IA by ClinicalTrials.gov. No research activities under NCT00670631 were conducted at IA. PRS staff have corresponded and neither party have data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No